CLINICAL TRIAL: NCT05564286
Title: Fosaprepitant Combined With Tropisetron Plus Dexamethasone in Preventing Nausea and Emesis During Fractionated Radiotherapy With Weekly Cisplatin Chemotherapy in Cervical Cancer and Nasopharyngeal Cancer
Brief Title: Triple Antiemetic Regimen for Chemoradiotherapy in Cervical Cancer or Nasopharyngeal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shantou University Medical College (Other)
Responsible Party: Principal Investigator, Chuangzhen Chen, Dr, Shantou University Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SUMC-Fosa
Record Dates: First submitted 2022-09-29; First posted 2022-10-03 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Cervical Cancer; Nasopharyngeal Cancer; Chemotherapy-induced Nausea and Vomiting; Radiation-Induced Nausea and Vomiting; Antiemetic
MeSH Terms: conditions — Uterine Cervical Neoplasms; Nasopharyngeal Neoplasms; Vomiting | interventions — fosaprepitant; Tropisetron; Dexamethasone

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- fosaprepitant group (Experimental): Intravenous fosaprepitant of 150mg was given before cisplatin administration on day 1. All patients received tropisetron 5mg and dexamethasone 5mg infusion on day 1 and oral dexamethasone 3.75 mg once a day on day 2-3.
  Interventions: Drug: Fosaprepitant; Drug: tropisetron; Drug: Dexamethasone
- control group (Active Comparator): The control group was delivered tropisetron 5mg and dexamethasone 5mg only.
  Interventions: Drug: tropisetron; Drug: Dexamethasone

INTERVENTIONS:
Drug: Fosaprepitant — In fosaprepitant group, patients would receive fosaprepitant combined with tropisetron plus dexamethasone to prevent chemoradiotherapy-induced nausea and vomitting while the control group would only be given tropisetron and dexamethasone .
  Other Names: shanqi
  Arms: fosaprepitant group
Drug: tropisetron — All patients received tropisetron 5mg on day 1.
  Other Names: luoting
Drug: Dexamethasone — .All patients received dexamethasone 5mg infusion on day 1 and oral dexamethasone 3.75 mg once a day on day 2-3.
  Other Names: xiluoan

SUMMARY:
The study is to evaluate the antiemetic effect of adding fosaprepitant to biplet regimen of tropisetron and dexamethasone for patients with cervical cancer or nasopharyngeal cancer treated with radiotherapy and concomitant weekly cisplatin chemotherapy in a south Chinese cohort.

DETAILED DESCRIPTION:
The study was designed as a prospective,randomized, single-blind control clinical trial aiming to assess the efficacy and safety of fosaprepitant combined with tropisetron and dexamethasone in preventing nausea and vomiting during 5 weeks of fractionated radiotherapy and concomitant weekly low-dose cisplatin chemotherapy in patients with cervical cancer or nasopharyngeal cancer.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed nasopharyngeal carcinoma (AJCC 8th stage II-IVa) or cervical cancer (adenocarcinoma, squamous cell carcinoma, or adenosquamous carcinoma, clinical FIGO stage Ib2-IVa;), planning to receive concurrent chemoradiotherapy),18 years or older, with an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.

Exclusion Criteria:

* took medications with antiemetic effect within 24 hours before initiation of concurrent chemoradiotherapy, had severe systemic diseases (such as uncontrolled diabetes/hypertension) or clinically unstable epileptic seizures require the use of anticonvulsants; allergic to fosaprepitant, tropisetron or dexamethasone.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
cumulative incidence of emesis overall phase | 5 weeks
  The primary endpoint of the study was the cumulative incidence of emesis overall phase (from 1st day of cycle 1 to 7th day of cycle 5, 7 days for one cycle).

CONTACTS AND LOCATIONS:
Overall Officials: Chuangzhen Chen, Principal Investigator — Shantou University Medical College
Locations (1):
- Cancer Hospital of Shantou University Medical College, Shantou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xie S, Huang R, Zhan Y, Cai Q, Wu Y, Huang K, Lin X, Wang R, Yan Y, Xie R, Wang S, Zeng C, Chen C. Efficacy of fosaprepitant combined with tropisetron plus dexamethasone in preventing nausea and emesis during fractionated radiotherapy with weekly cisplatin chemotherapy: interim analysis of a randomized, prospective, clinical trial using competing risk analysis. Support Care Cancer. 2023 Oct 18;31(12):640. doi: 10.1007/s00520-023-08111-9. PMID 37851143